CLINICAL TRIAL: NCT03163589
Title: Effect of Erythropoietin and Hypothermia on Management of Neonatal Hypoxic Ischemic Encephalopathy
Brief Title: Erythropoietin in Management of Neonatal Hypoxic Ischemic Encephalopathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ASAli, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHIE
Record Dates: First submitted 2017-05-18; First posted 2017-05-23 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Erythropoietin; Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Within 4 to 6 hours after birth all cases with moderate to severe hypoxic ischemic encephalopathy will be enrolled in therapeutic hypothermia using total body cooling and temperature and Receive erythropoietin (1000 U/kg intravenously) on days 1, 2, 3, 5 ,7 and 9 (six doses,first two doses will be daily from the first day and last 4 doses will be every 2 days)
  Interventions: Drug: Erythropoietin
- control group (Placebo Comparator): Within 4 to 6 hours after birth cases with moderate to severe hypoxic ischemic encephalopathy enrolled in therapeutic hypothermia using total body cooling and temperature and Receive normal saline on days 1, 2, 3, 5 ,7 and 9 (six doses,first two doses will be daily from the first day and last 4 doses will be every 2 days)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Erythropoietin — injection
  Arms: study group
Drug: normal saline — injection
  Arms: control group

SUMMARY:
Perinatal hypoxic-ischaemic encephalopathy occurs in one to three infants per 1000 term births, and up to 12 000 infants are affected each year in the united state of America. Hypoxic ischemic encephalopathy is not preventable in most cases, and therapies are limited. Hypothermia improves outcomes and is the current standard of care. Yet clinical trials suggest that 44% to 53% of infants who receive hypothermia will die or suffer moderate to severe neurological disability. Therefore, novel neuroprotective therapies are urgently needed to further reduce the rate and severity of neurodevelopmental disabilities resulting from hypoxic ischemic encephalopathy.

Erythropoietin is a novel neuroprotective agent, with remarkable neuroprotective and neuroregenerative effects in animals. Rodent and primate models of neonatal brain injury support the safety and efficacy of multiple erythropoietin doses for improving histological and functional outcomes after hypoxia-ischaemia.

DETAILED DESCRIPTION:
The cellular mechanisms by which erythropoietin exert neuroprotection are complex and not completely understood. In the acute period after hypoxia ischaemia, erythropoietin signaling in the brain induces several neuroprotective mechanisms. In addition to its anti-apoptotic and anti-inflammatory properties, erythropoietin also increases antioxidant activities and reduces excitotoxic cell injury.

In addition to its acute effects, erythropoietin stimulates growth factor release, enhances neurogenesis and angiogenesis, and promotes long-term repair and plasticity. Thus, erythropoietin provides neuroprotective and trophic effects that last well beyond the acute period of injury erythropoietin .enhances neurogenesis and directs multipotent neural stem cells to differentiate toward a neuronal cell fate.

In a clinical trial performed in China, Zhu et al. studied 167 neonates with of hypoxic ischemic encephalopathy that were randomized to receive erythropoietin (300-500U/kg) or placebo every second day for 2 weeks. The first dose of erythropoietin was given within 48 hours of delivery. Compared with placebo-treated infants, infants that received erythropoietin were less likely to die or have moderate to severe disability at 18 months of age (44% vs 25%, p=0.02).

Similarly, Elmahdy et al. studied 30 infants with hypoxic ischemic encephalopathy who were randomized to receive five daily doses of 2500 units/kg erythropoietin, or placebo, with the first dose given within 24 hours of delivery. The erythropoietin-treated infants demonstrated improved electroencephalography backgrounds, reduced biomarkers of oxidative stress after 2 weeks, and improved neurodevelopment at 6 months of age compared with placebo treated infants.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 36 weeks of gestational age.
2. whole body cooling within 6 hours after birth.
3. Perinatal depression based on at least one of the following:

   1. Apgar score < 5 at 10 minutes.
   2. Need for resuscitation at 10 minutes.
   3. pH < 7.1 in cord and Base deficit ≥ 15 mmol/L.
   4. Moderate or severe encephalopathy according to sernat and sernat staging.

Exclusion Criteria:

1-Admitted after 24 hour of birth. 2-Birth weight < 1800 g (e.g., intrauterine growth restriction) 3-Genetic or congenital condition that affects neurodevelopment. 3-Torch infection and neonatal sepsis. 4-complex congenital heart disease. 5-severe dysmorphic feature . 6-Microcephaly:Head circumference < 2 stander deviations below mean for gestational age.

7-Polycythemia (hematocrit > 65%). 8-Premature rupture of membrane or chorioamnionitis.

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Death or long-term major neurodevelopmental disability according to Griffith score. | 12 month
  The score is reported as normal if the score is between 85 and 114, mildly delayed if the score is 1 Stander deviation below the mean (<85), and significantly delayed if the score is 2 Stander deviation below the mean (<70)

SECONDARY OUTCOMES:
cerebral palsy | 12 month
  Presence and type of cerebral palsy determined using a standardized neurologic examination: no cerebral palsy,diplegic cerebral palsy,hemiplegic cerebral palsy, quadriplegic cerebral palsy.
Epilepsy. | 12 month age.
  define as 2 or more afebrile unprovoked seizure.
Magnetic resonance image evidence of brain injury. | 2-3 weeks after birth.
  The magnetic resonant imaging global scores will range from 48 to 186. score at 48 showing no evidence of acute injury; injury considers mild if the global score will between 49and 59, moderate if between 60 and 80 and severe if more than 81.
Electroencephalogram evidence of brain injury. | 1 weeks after birth
  EEG will be graded in to normal ,mild ,severe and isoelectric using EEG score according to Murray et al 2009
Adverse effect of erythropoietin | 12 months
  A-Hypertension: a systolic blood pressure in a neonate which is above 95th percentile for age and sex on three separate occasions; B- thrombotic events; C-polycythemia: central venous hematocrit of greater than 65%. D- red cell aplasia secondary to antierythropoietic antibodies. OR any other adverse effect appear during hospital stay or follow up.
seizure | during 2 weeks after birth
  number of clinical and electroencephalogram seizure

REFERENCES:
- [Background] Kurinczuk JJ, White-Koning M, Badawi N. Epidemiology of neonatal encephalopathy and hypoxic-ischaemic encephalopathy. Early Hum Dev. 2010 Jun;86(6):329-38. doi: 10.1016/j.earlhumdev.2010.05.010. Epub 2010 Jun 16. PMID 20554402
- [Background] Jacobs SE, Morley CJ, Inder TE, Stewart MJ, Smith KR, McNamara PJ, Wright IM, Kirpalani HM, Darlow BA, Doyle LW; Infant Cooling Evaluation Collaboration. Whole-body hypothermia for term and near-term newborns with hypoxic-ischemic encephalopathy: a randomized controlled trial. Arch Pediatr Adolesc Med. 2011 Aug;165(8):692-700. doi: 10.1001/archpediatrics.2011.43. Epub 2011 Apr 4. PMID 21464374
- [Background] Zacharias R, Schmidt M, Kny J, Sifringer M, Bercker S, Bittigau P, Buhrer C, Felderhoff-Muser U, Kerner T. Dose-dependent effects of erythropoietin in propofol anesthetized neonatal rats. Brain Res. 2010 Jul 9;1343:14-9. doi: 10.1016/j.brainres.2010.04.081. Epub 2010 May 7. PMID 20452333
- [Background] Zhu C, Kang W, Xu F, Cheng X, Zhang Z, Jia L, Ji L, Guo X, Xiong H, Simbruner G, Blomgren K, Wang X. Erythropoietin improved neurologic outcomes in newborns with hypoxic-ischemic encephalopathy. Pediatrics. 2009 Aug;124(2):e218-26. doi: 10.1542/peds.2008-3553. Epub 2009 Jul 27. PMID 19651565
- [Background] Elmahdy H, El-Mashad AR, El-Bahrawy H, El-Gohary T, El-Barbary A, Aly H. Human recombinant erythropoietin in asphyxia neonatorum: pilot trial. Pediatrics. 2010 May;125(5):e1135-42. doi: 10.1542/peds.2009-2268. Epub 2010 Apr 12. PMID 20385632
- [Background] Cirelli I, Bickle Graz M, Tolsa JF. Comparison of Griffiths-II and Bayley-II tests for the developmental assessment of high-risk infants. Infant Behav Dev. 2015 Nov;41:17-25. doi: 10.1016/j.infbeh.2015.06.004. Epub 2015 Aug 11. PMID 26276119
- [Background] Frymoyer A, Juul SE, Massaro AN, Bammler TK, Wu YW. High-dose erythropoietin population pharmacokinetics in neonates with hypoxic-ischemic encephalopathy receiving hypothermia. Pediatr Res. 2017 Jun;81(6):865-872. doi: 10.1038/pr.2017.15. Epub 2017 Jan 18. PMID 28099423
- [Background] Murray DM, Boylan GB, Ryan CA, Connolly S. Early EEG findings in hypoxic-ischemic encephalopathy predict outcomes at 2 years. Pediatrics. 2009 Sep;124(3):e459-67. doi: 10.1542/peds.2008-2190. Epub 2009 Aug 24. PMID 19706569
- [Background] Bednarek N, Mathur A, Inder T, Wilkinson J, Neil J, Shimony J. Impact of therapeutic hypothermia on MRI diffusion changes in neonatal encephalopathy. Neurology. 2012 May 1;78(18):1420-7. doi: 10.1212/WNL.0b013e318253d589. Epub 2012 Apr 18. PMID 22517107